CLINICAL TRIAL: NCT07291037
Title: A Phase III, Randomised, Open-Label, Multicentre Study of Datopotamab Deruxtecan or Docetaxel in Previously Treated TROP2-positive Advanced or Metastatic Non-squamous Non-Small Cell Lung Cancer Without Actionable Genomic Alterations (TROPION-Lung17)
Brief Title: Phase III Study of Datopotamab Deruxtecan Versus Docetaxel in Previously Treated TROP2-positive Advanced or Metastatic Non-squamous NSCLC Without Actionable Genomic Alterations
Acronym: TROPION-Lung17
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D763QC00001; 2024-520101-39-00 (Other: EU CT Number)
Record Dates: First submitted 2025-10-28; First posted 2025-12-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: TROPION-Lung17; Non-small cell lung cancer (NSCLC); Advanced non-squamous NSCLC; Metastatic non-squamous NSCLC; Datopotamab deruxtecan (Dato-DXd; DS-1062a); Docetaxel; Trophoblast cell surface protein 2 (TROP2); Normalised membrane ratio (NMR)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: Arm A: Datopotamab deruxtecan monotherapy
  Arm B: Docetaxel monotherapy
Masking Description: TROPION-Lung17 is an open-label study; however, the study will be conducted as 'Sponsor-blind'.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Datopotamab deruxtecan (Dato-DXd) monotherapy (Experimental): Participants in the Dato-DXd monotherapy group will receive Dato-DXd as intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Interventions: Drug: Datopotamab deruxtecan (Dato-DXd)
- Arm B: Docetaxel monotherapy (Active Comparator): Participants in the docetaxel monotherapy group will receive docetaxel as intravenous (IV) infusion every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Datopotamab deruxtecan (Dato-DXd) — Dato-DXd administered intravenously (IV)
  Other Names: DS-1062a
  Arms: Arm A: Datopotamab deruxtecan (Dato-DXd) monotherapy
Drug: Docetaxel — Docetaxel administered intravenously (IV)
  Arms: Arm B: Docetaxel monotherapy

SUMMARY:
TROPION-Lung17 will measure the efficacy and safety of datopotamab deruxtecan (Dato-DXd) compared with docetaxel in patients with trophoblast cell surface protein 2 (TROP2) positive advanced or metastatic lung cancer without actionable genomic alterations (AGA).

DETAILED DESCRIPTION:
TROPION-Lung17 is a phase III, 2-arm, randomised, open-label, multicentre study, assessing the efficacy and safety of Dato-DXd compared with docetaxel in participants with previously treated trophoblast cell surface protein 2 (TROP2) normalised membrane ratio (NMR) positive advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) without actionable genomic alterations (AGA), and to assess the clinical performance of the investigational in vitro diagnostic (IVD) device.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented Stage IIIB, IIIC, or Stage IV non-squamous non-small cell lung cancer (NSCLC) without actionable genomic alterations (AGA) at the time of randomisation and meets the criteria for NSCLC:

  * Participants must have documented negative test results for epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), and ROS proto-oncogene 1 (ROS1) genomic alterations.
  * Has no known tumour genomic alterations in neurotrophic tyrosine receptor kinase (NTRK), proto-oncogene B-raf (BRAF), rearranged during transfection (RET), mesenchymal-epithelial transition (MET) exon 14 skipping, Kirsten rat sarcoma viral oncogene homolog (KRAS) G12C, human epidermal growth factor receptor 2 (HER2) or any other actionable driver oncogenes for which there are locally approved and available targeted first-line therapies.
  * Prospectively assessed trophoblast cell surface protein 2 (TROP2) normalised membrane ratio (NMR) positive.
* Documentation of radiographic disease progression while on or after receiving the most recent treatment regimen for advanced or metastatic NSCLC.
* Participants must have received platinum based chemotherapy (PBC) in combination with anti-programmed death-protein 1 (anti-PD-1)/anti-programmed death-ligand 1 (anti-PD-L1) monoclonal antibody (mAb) as the only prior line of therapy or received PBC and anti-PD-1/anti-PD-L1 monoclonal antibody (in either order) sequentially as the only 2 prior lines of therapy.
* Provision of acceptable formalin fixed and paraffin embedded (FFPE) tumour sample for assessment of TROP2.
* At least one lesion not previously irradiated that qualifies as a Response Evaluation Criteria in Solid Tumours, Version 1.1 (RECIST 1.1) target lesion (TL) at baseline and can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and is suitable for accurate repeated measurements.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* Adequate bone marrow reserve and organ function within 7 days before randomisation.

Exclusion Criteria:

* Squamous, mixed NSCLC, or small cell lung cancer (SCLC) histology.
* NSCLC disease that is eligible for definitive local therapy alone.
* History of another primary malignancy other than NSCLC, except for malignancy treated with curative intent with no known active disease within 3 years before randomisation and of low potential risk for recurrence.
* Spinal cord compression or brain metastases, unless asymptomatic, stable, and not requiring treatment with corticosteroids or anticonvulsants for at least 7 days prior to randomisation.
* Clinically significant corneal disease.
* Has active or uncontrolled hepatitis B or C virus infection.
* Known human immunodeficiency virus (HIV) infection that is not well controlled.
* Uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals.
* History of non-infectious interstitial lung disease (ILD)/pneumonitis including radiation pneumonitis that required steroids, has current ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
* Severe pulmonary function compromise per Investigator discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2029-01-29 (Estimated); Study Completion 2029-01-29 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 2.5 years
  PFS is defined as the time from randomization until radiological progression per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) as assessed by Blinded Independent Central Review (BICR), or death due to any cause.
Overall survival (OS) | Approximately 3.5 years
  OS is defined as the time from randomization until the date of death due to any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 2.5 years
  ORR is defined as the proportion of participants who have a confirmed complete response (CR) or confirmed partial response (PR), as determined by Blinded Independent Central Review (BICR) per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1).
Duration of response (DoR) | Approximately 2.5 years
  DoR is defined as the time from the date of first documented response until the date of documented progression per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1), as assessed by Blinded Independent Central Review (BICR) or death due to any cause.
Time to second progression or death (PFS2) | Approximately 2.5 years
  PFS2 is defined as the time from randomization until the earliest of the progression event (following the initial progression event), after first subsequent therapy, or death. The date of the second progression will be recorded by the Investigator in the electronic Case Report Form (eCRF) and defined according to local standard clinical practice based on radiological or clinical progression.
Exposure-efficacy relationship | Approximately 2.5 years
  Evaluate the relationship between plasma concentrations of Dato-DXd (µg/mL) and efficacy endpoints (PFS, OS), as evaluated by cox-proportional hazard model.
Exposure-safety relationship | Approximately 2.5 years
  Evaluate the correlation between concentrations of Dato-DXd (µg/mL) and safety endpoints (including Gr3+AE, AESIs), as evaluated by logistic regression
Covariates effect on exposure | Approximately 2.5 years
  Evaluate the relationship between covariates (including but not limited to age, sex, body weight, race) and plasma concentrations of Dato-DXd (µg/mL) and/or DXd (ng/mL), as evaluated by population PK model
Immunogenicity of datopotamab deruxtecan (Dato-DXd) | Approximately 2.5 years
  Presence of antidrug antibodies (ADAs) for Dato-DXd.
Participant-reported lung cancer symptoms of non-small cell lung cancer (NSCLC) | Approximately 2.5 years
  Time to deterioration (TTD) in pulmonary symptoms (dyspnoea, cough, and chest pain) as measured by the Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ).
  Scores range from a minimum of 0 to a maximum of 20, with higher scores indicating more symptom burden.
  TTD is defined as time from randomization to the date of first deterioration.
  Deterioration is defined as change from baseline that reaches an meaningful change threshold (MCT).
Participant-reported physical functioning | Approximately 2.5 years
  Time to deterioration (TTD) in physical functioning as measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form - Physical Function 8c.
  TTD is defined as time from randomization to the date of first deterioration.
  Deterioration is defined as change from baseline that reaches a meaningful change threshold (MCT).
Participant-reported global health status (GHS)/quality of life (QoL) | Approximately 2.5 years
  Time to deterioration (TTD) in GHS/QoL as measured by the European Organization for Research and Treatment of Cancer Item Library 172 (EORTC IL172).
  Scores range from a minimum of 0 to a maximum of 100, with higher scores indicating a better outcome.
  TTD is defined as time from the date of randomisation to the date of first deterioration.
  Deterioration is defined as change from baseline that reaches a meaningful change threshold (MCT).
Correlation of TROP2 expression at various cut offs with clinical response | Approximately 2.5 years
  Evaluate the relationship between TROP2 NMR expression and efficacy endpoints.
Diagnostic development and biomarker assay concordance analysis | Approximately 2.5 years
  Evaluate the relationship between TROP2 NMR status at a defined cutoff and efficacy endpoints, as determined by the diagnostic device.

CONTACTS AND LOCATIONS:
Locations (173):
- United States (49):
  - Research Site, Chandler, Arizona
  - Research Site, Gilbert, Arizona
  - Research Site, Goodyear, Arizona
  - Research Site, Duarte, California
  - Research Site, Irvine, California
  - Research Site, La Jolla, California
  - Research Site, Loma Linda, California
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, Grand Junction, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Newnan, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Niles, Illinois
  - Research Site, Zion, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, South Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Brandywine, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Bridgeton, Missouri
  - Research Site, Columbia, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Albuquerque, New Mexico
  - Research Site, East Syracuse, New York
  - Research Site, Portland, Oregon
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Denton, Texas
  - Research Site, Plano, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Williamsburg, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Eau Claire, Wisconsin
- Australia (5):
  - Research Site, Gosford
  - Research Site, Kogarah
  - Research Site, South Brisbane
  - Research Site, St Albans
  - Research Site, Wollongong
- Austria (4):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Rankweil
  - Research Site, Vienna
- Belgium (5):
  - Research Site, Hasselt
  - Research Site, La Louvière
  - Research Site, Libramont-Chevigny
  - Research Site, Namur
  - Research Site, Sint-Niklaas
- Brazil (3):
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (6):
  - Research Site, Vancouver, British Columbia
  - Research Site, Moncton, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
- China (21):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jiamusi
  - Research Site, Jinan
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xuzhou
  - Research Site, Zhengzhou
- Germany (15):
  - Research Site, Bad Saarow
  - Research Site, Bielefeld
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Krefeld
  - Research Site, Minden
  - Research Site, Oldenburg
  - Research Site, Troisdorf
  - Research Site, Velbert
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Törökbálint
- India (5):
  - Research Site, Bangalore
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Nashik
  - Research Site, New Delhi
- Italy (5):
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Rozzano
- Japan (15):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Iwakuni-shi
  - Research Site, Kashiwa
  - Research Site, Kawasaki-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Poland (4):
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
- South Korea (4):
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (7):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Zaragoza
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Muang
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Istanbul
- United Kingdom (5):
  - Research Site, Huddersfield
  - Research Site, London
  - Research Site, Maidstone
  - Research Site, Norwich
  - Research Site, Stoke-on-Trent
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca (AZ) group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for Important Protocol Deviation (IPD), but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the European Federation of Pharmaceutical Industries and Associations (EFPIA)/Pharmaceutical Research and Manufacturers of America (PhRMA) Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/